CLINICAL TRIAL: NCT01349764
Title: Effect of Vitamin D Replacement in Vitamin D Deficient Patients With History of Urolithiasis: A Randomized Controlled Trial
Brief Title: Effect of Vitamin D Replacement in Patients With Urolithiasis
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit required sample size
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr Sero Andonian, Associate Professor of Urology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 10-325-BMB
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Urolithiasis
Keywords: vitamin D replacement; Urolithiasis; deficiency; insufficiency
MeSH Terms: conditions — Urolithiasis | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No vitamin D replacement: The control arm will not receive vitamin D replacement, but patients in both study arms will receive care consistent with best care practices for stone disease. All patients will be evaluated by the stone clinic clinical nutritionist and full nutritional evaluation will be performed. All patients will be advised to maintain adequate hydration (>2L/day), no-added salt diet (Na 80-100mmol/day), low protein diet (1 g/kg/day). Patients with hyperoxaluria will be advised to follow low-oxalate diet. All patients will be advised to maintain moderate calcium intake; 800-1200mg/day.
- Vitamin D3 tabs: The active arm of randomization will receive vitamin D repletion in the form of oral vitamin D3 tablets 10 000 IU twice/ week for 8 consecutive weeks, followed by a maintenance dose of 1 000 IU daily for further 22 months.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3
  Groups: Vitamin D3 tabs

SUMMARY:
When Vitamin D replacement is initiated in patients with history of urolithiasis, there will be higher incidence of hypercalciuria but with careful follow-up of these patients, hypercalciuria could be appropriately managed with thiazide diuretics so that the risk of newly diagnosed renal stones will be equivalent to control groups without Vitamin D replacements.the purpose of the study is to determine the effect of vitamin D replacement in patients with previous history of urolithiasis presenting to a tertiary stone clinic in terms of changes in 24-hour urine collection parameters and to evaluate the lithogenic effect of vitamin D replacement in terms of development of urolithiasis. Eighty-six eligible patients will be included in terms of having suboptimal vitamin D with history of calcareous urolithiasis and urinary calcium excretion <7.5 mmol/day. Patients will be randomly divided into 2 equal groups depending on whether they will receive vitamin D replacement with follow-up at 3, 6, 12, & 24 months.

DETAILED DESCRIPTION:
During the last year, clinical studies on vitamin D have confirmed the presence of world-wide incidence of vitamin D deficiency. Recently, the investigators detected an incidence of 80% vitamin D deficiency/ insufficiency in patients presenting to our tertiary stone clinic. However, there is no data in the literature regarding the safety of vitamin D replacement in this highly specialized group of patients. Consequently, clinicians are concerned about vitamin D replacement in these patients for fear of increased risk of hypercalciuria and stone formation.

This study aims to determine the effect of vitamin D replacement on patients presenting to a tertiary stone clinic in terms of changes in 24-hour urine collection parameters and secondary stone formation. Eighty- six eligible patients with 25-(OH)D deficiency or insufficiency (defined as serum level <72 nmol/L) with history of calcareous urolithiasis and urinary calcium excretion <7.5 mmol/day will be included in the study.

Eligible patients will be randomly divided into 2 equal groups depending on whether they will receive vitamin D replacement or not. Randomization will be done using a computer-based random number generator. Patients will receive vitamin D3 tablets 10.000 IU twice a week for 8 weeks followed by a maintenance dose of 1.000 IU daily for 21 months. All patients will be subjected to full history taking and clinical examinations, urinalysis and culture when indicated, liver function tests, urea and creatinine, ionized normalized calcium, phosphate, magnesium, uric acid, potassium, PTH, TSH and both forms of vitamin D [25(OH)D and 1, 25 (OH)2D], low dose CT scan to confirm stone free status and baseline bone density scan, together with metabolic stone workup consisting of stone analysis and two 24-hour urine collections for calculation of volume, osmolality, pH, creatinine, urea, calcium, phosphate, chloride, magnesium, sodium, potassium, oxalate, citrate, uric acid, and quantitative cystine. Similar follow-up measures will be done at 3, 6, 12, 18 & 24 months. At the end of the study, low dose CT scan and bone density scans will be repeated.

Data will be collected and tabulated using the commercially available SPSS software version 17 (SPSSInc, Chicago, IL, USA). Descriptive statistics will be presented in terms of percentage, frequency, means and standard deviations for parametric variables and median with interquartile ranges for non-parametric. Differences between both groups will be compared with the Fisher's exact test for categorical data and Student's t- test for the continuous variables. In addition, interplay of more than 2 variables will be analysed using multivariate logistic-regression. The effect of season of recruitment on and changes in serum 25(OH)D will be evaluated using multivariate analysis of covariance (ANCOVA) with two-tailed p-values less than values 0.05 representing statistical significance. Time to hypercalciuria or time to stone formation c will be analysed using a survival analysis technique and comparison of the 2 groups using a log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* 25-OHD deficiency or insufficiency (defined as serum level <75 nmol/L).
* History of urolithiasis (Calcareous stones).
* 24-hour urinary calcium excretion <7.5 mmol/day (normocalciuric).
* Low fracture risk (estimated by FRAX®, which was developed by WHO).

Exclusion Criteria:

* Age < 18 years
* Renal dysfunction (Serum creatinine concentrations of > 150 μmol/L).
* History of non-calcareous stones e.g. uric acid, cystine, or struvite stones.
* Hypercalcemia (serum ionized normalized calcium > 1.32 mmol/L)
* Patients with secondary hypercalciuria e.g. primary hyperparathyroidism, sarcoidosis, hyperthyroidism, or active malignancy.
* Evidence of osteoporosis or intermediate/high fracture risk (estimated by FRAX).
* Patients taking drugs that could potentially affect urinary calcium excretion (vitamin D, calcium supplement, loop diuretics, steroids, or lithium).
* Evidence of liver dysfunction or other disorders that may cause non-nutritional vitamin D deficiency or abnormal bone development.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the MUHC stone clinic and had inadequate vitamin D.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The effect of vitamin D replacement in patients with previous history of urolithiasis presenting to a tertiary stone clinic in terms of changes in 24-hour urine collection parameters | 6 months

SECONDARY OUTCOMES:
The lithogenic effect of vitamin D replacement in terms of development of urolithiasis. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sero Andonian, MD, FRCS (C), Principal Investigator — MUHC, Montreal QC, Canada; Ahsan Alam, MD, FRCP (C), Study Director — MUHC, Montreal QC, Canada; Ramsey Sabbagh, MD, FRCP (C), Study Director — MUHC, Montreal QC, Canada; Bernard Unikowsky, MD, FRCP (C), Study Director — MUHC, Montreal QC, Canada
Locations (1):
- Royal Victoria Hospital, McGill University Health Center, Montreal, Quebec, Canada